CLINICAL TRIAL: NCT02248883
Title: Assessment of Electrophysiological Effects of Tipranavir Co-administered With Ritonavir Given b.i.d. for 2.5 Days on the QT Interval in Healthy Female and Male Subjects. A Double-blind, Randomised, Placebo Controlled, Two-way Crossover Study With a Positive Control (Moxifloxacin) and Parallel Dose Groups
Brief Title: Electrophysiological Effects of Tipranavir Co-administered With Ritonavir on the QT Interval in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1182.60
Record Dates: First submitted 2014-09-24; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

ARMS (3):
- low TPV/RTV (Experimental)
  Interventions: Drug: TPV low; Drug: Moxifloxacin; Drug: RTV
- high TPV/RTV (Experimental)
  Interventions: Drug: Moxifloxacin; Drug: TPV high; Drug: RTV
- Placebo/RTV (Experimental)
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: RTV

INTERVENTIONS:
Drug: TPV low
  Arms: low TPV/RTV
Drug: Placebo
  Arms: Placebo/RTV
Drug: Moxifloxacin
  Other Names: Avelox®
Drug: TPV high
  Arms: high TPV/RTV
Drug: RTV

SUMMARY:
To demonstrate that tipranavir (TPV) co-administered with ritonavir (RTV) does not affect the QT interval more than placebo co-administered with ritonavir

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male volunteers as determined by the results of screening according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
2. Age ≥ 18 and Age ≤ 55 years
3. BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Gastrointestinal tract surgery (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts.
5. Relevant acute, chronic or active chronic infections (e.g. hepatitis, HIV).
6. History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Smoker (more than 10 cigarettes/day or 3 cigars/day or 3 pipes/day)
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Veins unsuited for i.v. puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. History of any bleeding disorder or acute blood coagulation defect
17. Hypersensitivity to ritonavir, moxifloxacin and/or related drugs of these classes
18. History of Glucose-6-phosphate-deficiency
19. Excessive physical activities (within one week prior to trial or during the trial)
20. Any laboratory value outside the reference range that is of clinical relevance
21. A history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
22. Heart rate at screening of > 80 bpm or < 45 bpm
23. Any screening ECG value outside of the reference range of clinical relevance including, but not limited to PR interval > 240 ms, QRS interval > 120 ms, QTcB or QTcF > 450 ms, or QT (uncorrected) > 470 ms
24. Inability to comply with the dietary regimen of the study centre

    For female subjects:
25. Pregnancy
26. Positive pregnancy test
27. No adequate contraception (adequate contraception e.g. sterilisation, intrauterine pessary (IUP) or oral contraception not containing ethinyl estradiol)
28. Oral contraception containing ethinyl estradiol without the use of an additional barrier method
29. Hormone replacement containing ethinyl estradiol
30. Inability to maintain this adequate contraception during the whole study period
31. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2005-12; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in individually heart rate corrected QT interval length (QTcI) | baseline and 2 to 4 hours after drug administration on day3

SECONDARY OUTCOMES:
Change from baseline in (QTcI) | baseline and 2 to 4 hours after drug administration on day 1
Change from baseline in (QTcI) | baseline and 1 to 12 hours after drug administration on day1 and 3